CLINICAL TRIAL: NCT06901011
Title: Continuous Renal Replacement Therapy Doses in Critically Ill Patients With Acute Kidney Injury
Acronym: CRRIT1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Hospital Clinic i provincial de Barcelona (Unknown)
Responsible Party: Principal Investigator, Fritz Diekmann, Research Coordinator of the Institute of Nephrology and Urology (ICNU) at Hospital Clínic de Barcelona, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2024/0228
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-03

CONDITIONS: Renal Replacement Therapy for Acute Kidney Injury in ICU; Continuous Renal Replacement Therapy (CRRT)
Keywords: Continuous Renal Replacement Therapy (CRRT); Renal Replacement Therapy for Acute Kidney Injury in ICU; dialytrauma
MeSH Terms: interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Intervention Model Description: Prospective comparative intervention study, Single-center. Randomized, open-label study
Masking Description: Statistical analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Effluent dose schedule of 10-20 ml/kg/h after 48 hours of starting dose of 25-35 ml/kg/h, until completing 96 hours
  Interventions: Procedure: continuous renal replacement therapy
- Control (No Intervention): Effluent dosage schedule of 25-35 ml/kg/h fixed for 96 hours

INTERVENTIONS:
Procedure: continuous renal replacement therapy — Intervention Arm: Effluent dose schedule of 10-20 ml/kg/h after 48 hours of starting dose of 25-35 ml/kg/h, until completing 96 hours
  Control Arm Effluent dosage schedule of 25-35 ml/kg/h fixed for 96 hours
  Other Names: continuous renal replacement dose
  Arms: Intervention

SUMMARY:
Acute kidney injury in critically ill patients admitted to the ICU is a common complication associated with high mortality or long-term chronic kidney damage. Some of these patients require continuous renal replacement therapy (low-intensity hemodialysis for 24 hours) until renal function recovery is achieved.

Continuous Renal Replacement Therapy (CRRT) is a crucial treatment for ICU patients with acute renal failure. It offers continuous toxin removal and prevents fluid accumulation in the patient's body. The therapy not only eliminates toxins but also physiological substances, including micronutrients and essential elements for cellular metabolism and organ function.

Currently, there is limited information available to adjust the renal therapy dose and avoid or balance the loss of these substances without causing toxin accumulation. Some studies suggest that high doses of therapy do not provide benefits and increase complications.

The objective of this study is to evaluate two doses of continuous renal therapy in terms of internal environment control (sodium, potassium, and acids and bases), micronutrient loss, and toxin elimination. After 48 hours of therapy, patients will be assigned to continue with a dose equal to the initial dose or a decrease in the initial dose. These two options are part of the current standard practice in our center.

Patients participating in the study will be randomly assigned one of the continuous renal therapy doses. The study is open, so treating physicians will always know the therapy the patient is receiving and can freely adjust it if deemed necessary.

The intervention duration is 96 hours, after which the dose will be at the discretion of the treating medical team. A follow-up will be conducted through medical records or phone calls approximately 90 days after starting therapy.

The risks for the patient are minimal, as toxin elimination monitoring will be even more intensive than usual. The study plans to include approximately 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Acute renal failure (AKIN 3) requiring Continuous Renal Replacement Therapy
* Requirement of vasoactive drugs (norepinephrine > 0.1 mcg/kg/min)
* Written informed consent (patient or family)

Exclusion Criteria:

* Lack of informed consent.
* Possibility of using plasma exchange or MARS therapy at the at the time of inclusion.
* Baseline renal function with an estimated glomerular filtration rate (CKD-EPI) less than 30 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Control of biochemical parameters (natremia, kalemia, and base excess) | From enrollment to the end of follow-up at 90 days
  To compare the impact of a reduced dose of effluent regimen in CRRT (10-20 ml/kg/h), after 48 hours of 25-35 ml/kg/h dose, on the control of internal homeostasis parameters (Natremia, kalemia and base excess) compared to a fixed dose of 25-35 ml/kg/h for 96 hours of CRRT.

CONTACTS AND LOCATIONS:
Overall Officials: Gaston J Piñeiro, MD, PhD, Principal Investigator — Hospital Clínic of Barcelona

IPD SHARING:
Plan to Share IPD: Undecided
The sharing of participants' individual data with third parties must be evaluated by the center's Research Ethics Committee. Collection of individual data may only be carried out within the parameters permitted by European data protection legislation.

REFERENCES:
- [Background] Koekkoek KWA, Berger MM. An update on essential micronutrients in critical illness. Curr Opin Crit Care. 2023 Aug 1;29(4):315-329. doi: 10.1097/MCC.0000000000001062. Epub 2023 Jun 8. PMID 37306546
- [Background] Karkar A, Ronco C. Prescription of CRRT: a pathway to optimize therapy. Ann Intensive Care. 2020 Mar 6;10(1):32. doi: 10.1186/s13613-020-0648-y. PMID 32144519
- [Background] Fayad AI, Buamscha DG, Ciapponi A. Intensity of continuous renal replacement therapy for acute kidney injury. Cochrane Database Syst Rev. 2016 Oct 4;10(10):CD010613. doi: 10.1002/14651858.CD010613.pub2. PMID 27699760
- [Background] Jun M, Heerspink HJ, Ninomiya T, Gallagher M, Bellomo R, Myburgh J, Finfer S, Palevsky PM, Kellum JA, Perkovic V, Cass A. Intensities of renal replacement therapy in acute kidney injury: a systematic review and meta-analysis. Clin J Am Soc Nephrol. 2010 Jun;5(6):956-63. doi: 10.2215/CJN.09111209. Epub 2010 Apr 15. PMID 20395356
- [Background] RENAL Replacement Therapy Study Investigators; Bellomo R, Cass A, Cole L, Finfer S, Gallagher M, Lo S, McArthur C, McGuinness S, Myburgh J, Norton R, Scheinkestel C, Su S. Intensity of continuous renal-replacement therapy in critically ill patients. N Engl J Med. 2009 Oct 22;361(17):1627-38. doi: 10.1056/NEJMoa0902413. PMID 19846848
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Maynar Moliner J, Honore PM, Sanchez-Izquierdo Riera JA, Herrera Gutierrez M, Spapen HD. Handling continuous renal replacement therapy-related adverse effects in intensive care unit patients: the dialytrauma concept. Blood Purif. 2012;34(2):177-85. doi: 10.1159/000342064. Epub 2012 Oct 24. PMID 23095418
- [Background] Chawla LS. Permissive azotemia during acute kidney injury enables more rapid renal recovery and less renal fibrosis: a hypothesis and clinical development plan. Crit Care. 2022 Apr 28;26(1):116. doi: 10.1186/s13054-022-03988-0. PMID 35484549